CLINICAL TRIAL: NCT05692830
Title: Towards a Wearable Alcohol Biosensor: Examining the Accuracy of BAC Estimates From New-Generation Transdermal Technology Using Large-Scale Human Testing and Machine Learning Algorithms
Status: Recruiting | Type: Observational
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Catharine Fairbairn, Associate Professor, University of Illinois at Urbana-Champaign
Other Study IDs: AA028488-01A1
Record Dates: First submitted 2022-10-20; First posted 2023-01-20 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Drinking; Alcohol Intoxication
Keywords: transdermal alcohol content; ambulatory; transdermal biosensor; machine learning algorithms; breath alcohol content
MeSH Terms: conditions — Alcohol Drinking; Alcoholic Intoxication | interventions — Ethanol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Alcohol — Alcohol administered orally at multiple doses and consumption speeds to test transdermal device accuracy

SUMMARY:
The study will employ a combined laboratory-ambulatory design. Participants will engage in ambulatory assessment over the course of 14 days, wearing biosensors assessing transdermal alcohol concentration (TAC) and providing breathalyzer readings in real-world contexts. Also during this period, participants will attend three laboratory alcohol-administration sessions scheduled at one-week intervals, with alcohol dose and rate of consumption manipulated within and between participants, respectively. Laboratory visits will also double as ambulatory orientation, check-in, and close-out sessions.

DETAILED DESCRIPTION:
Laboratory Procedures: The aim of the laboratory study is to capture variability in the TAC-BAC relationship across individuals in a controlled context, featuring manipulations theorized to confound transdermal measurements of BAC and so ensuring adequate variability in these factors in the broader dataset. Laboratory alcohol-administration sessions will be held at one-week intervals, scheduled at study initiation (day 0), study midpoint (day 7), and study end (day 14).

Alcohol-administration procedures will employ a within (alcohol dose) X between (rate of consumption) participant design. All participants will consume three doses of alcohol over the course of the three laboratory sessions, targeting peak blood alcohol concentration (BAC) levels of .03%, .06%, and .09% respectively. The order of alcohol doses will be counterbalanced across participants. The exact quantity of alcohol administered to each participant in order to achieve these target peak BACs will be calculated based on individualized formulas adjusting for drinking rate, sex, height, weight, and age (see formulas provided in Watson et al., (1981)). Rate of consumption will be manipulated between participants, with equal numbers of participants assigned to consume alcohol at relatively "fast" and "slow" rates. Beverage intake will be monitored to ensure participant comfort and even consumption across the beverage administration period. After beverage administration, participants will provide breath alcohol concentration (BrAC) readings at 10- min intervals.

In addition, during the laboratory procedures, participants will be exposed to environmental factors that are known to impact readings taken by transdermal sensors. These manipulations will allow the research team to train the machine learning algorithm to recognize and model for these environmental effects. These manipulations include: 1) Environmental alcohol: common household products containing alcohol (e.g., hand sanitizer, perfume, lotion containing alcohol) will be sprayed or applied in proximity to the transdermal sensor; 2) Sweating: Participants will be asked to engage in a brief 10-30 minute aerobic exercise while in a seated position (i.e., stationary biking) while under the supervision of a research assistant. This brief exercise will be designed simply to yield exertion to the point of sweating and not exertion beyond this point; 3) Arm Movements: Participants will be asked to engage in isolated body movements (e.g., arms and feet) to determine whether device shifting caused by such movements impact readings taken by transdermal sensors.

Ambulatory Procedures: This arm of the study aims to capture the TAC-BAC relationship among participants drinking in everyday settings. Ambulatory assessment will take place over 14 days. During laboratory session 1, prior to beverage administration, participants will be oriented to ambulatory study procedures. One or more transdermal device will be worn throughout participation. During orientation, participants will be trained to use the mobile breathalyzer. To avoid contamination of breathalyzer readings by mouth alcohol, participants will be instructed to wait 5 minutes after their last sip of alcohol to provide a reading. Also during this orientation session, participants will receive training in standard drink reporting (used to validate breathalyzer readings). During ambulatory assessment, participants will provide breathalyzer readings in response to both random and user-initiated prompts via their smartphones. On day 14 of the study, participants will attend a final laboratory session during which they will return study equipment as well as complete questionnaires asking them to reflect on their experience using the transdermal sensors and their likelihood to adopt a transdermal sensor application.

Since initial record creation, the study start date has been updated to conform to current ICMJE pre-registration requirements. Only participants recruited subsequent, and not prior to, this updated initiation date are included in reports from the main trial.

ELIGIBILITY:
Inclusion Criteria:

* 21 years or older
* drink alcohol at least 2x weekly

Exclusion Criteria:

* psychological or medical conditions that might contraindicate alcohol-administration
* history of adverse reaction to type and amount of beverage used in the study
* currently seeking treatment for alcohol use disorder
* does not drink alcohol regularly
* taking drugs or medications for which alcohol consumption would be contraindicated
* women who are pregnant or are attempting to become pregnant

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Regular healthy drinkers aged 21+
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-10-22 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Transdermal estimates of alcohol consumption | Across the 14 day period of the study
  We will assess the accuracy of transdermal estimates of drinking vs sobriety
Transdermal estimates of drinking risk level | Across the 14 day period of the study
  We will assess the accuracy of transdermal estimates of high risk drinking vs low risk drinking and sobriety
Transdermal estimates of blood alcohol concentration | Across the 14 day period of the study
  We will assess the accuracy of transdermal estimates of blood alcohol concentration (BAC)

CONTACTS AND LOCATIONS:
Overall Officials: Catharine Fairbairn, PhD, Principal Investigator — University of Illinois Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Champaign, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kornacki B, Szreterowa M, Jablonska-Budajowa U, Goryszewska-Maciochowa H. [Transciliary lensectomy]. Klin Oczna. 1983 Nov-Dec;85(11-12):421-3. No abstract available. Polish. PMID 6668891
- [Background] Bragg DG. Radiologic manpower. Issues and controversies. Invest Radiol. 1987 Jun;22(6):515. doi: 10.1097/00004424-198706000-00015. No abstract available. PMID 3623856
- [Background] Leemhuis MP, Blom PS, Koevoet A. [Beta-carotene loading test as a screening test for steatorrhea]. Ned Tijdschr Geneeskd. 1971 Sep 11;115(37):1527-30. No abstract available. Dutch. PMID 5569301
- [Background] Haxby DG, Rodriguez GS, Zechnich AD, Schuff RA, Tanigawa JS. Manufacturers' distribution of drug samples to a family medicine clinic. Am J Health Syst Pharm. 1995 Mar 1;52(5):496-9. doi: 10.1093/ajhp/52.5.496. PMID 7606553
- [Background] Graham-Pole J. Treating acute lymphoblastic leukaemia after relapse: bone marrow transplantation or not? Lancet. 1989 Dec 23-30;2(8678-8679):1517-8. doi: 10.1016/s0140-6736(89)92953-x. No abstract available. PMID 2574782
- [Background] Murdaugh HV Jr, Robin ED, Millen JE, Drewry WF, Weiss E. Adaptations to diving in the harbor seal: cardiac output during diving. Am J Physiol. 1966 Jan;210(1):176-80. doi: 10.1152/ajplegacy.1966.210.1.176. No abstract available. PMID 5323319
- [Background] Lange DE. [Use of antibiotics in periodontal problem cases for prevention of bacteremia and prophylaxis of bacterial endocarditis]. Quintessenz. 1988 Jun;39(6):1047-51. No abstract available. German. PMID 3217504
- [Background] Griesbach WE, Chaikoff IL, Nichols CW Jr, Goldberg RC. Formation of adenomata in hypophyses of rats subjected to both subtotal thyroidectomy and administration of 131-I, and its prevention by feeding of desiccated thyroid. Cancer Res. 1965 Nov;25(10):1804-16. No abstract available. PMID 4159387
- [Background] Vihma Y, Korppi-Tommola T, Parkkulainen KV. Pelviureteric obstruction in children: the effect of pyeloplasty on 99mTc-DTPA uptake and washout. Z Kinderchir. 1984 Dec;39(6):358-63. doi: 10.1055/s-2008-1044245. PMID 6395541
- [Background] Martelli MF, Falini B, Tabilio A, Aversa F. Topographical localization of intracellular immunoglobulins in hairy cells by immunoelectron microscopy. Acta Haematol. 1980;64(5):251-5. doi: 10.1159/000207277. PMID 6779481
- [Background] Van Iddekinge B. Ectopic pregnancy: a review. S Afr Med J. 1972 Nov 25;46(47):1844-9. No abstract available. PMID 4265311
- [Background] Molthan L, Crawford MN. Three examples of anti-Lub and related data. Transfusion. 1966 Nov-Dec;6(6):584-9. doi: 10.1111/j.1537-2995.1966.tb04782.x. No abstract available. PMID 5951618
- [Background] Kopysc Z, Barczyk K, Krol E. [A new syndrome in the group of euhydrotic ectodermal dysplasias]. Pediatr Pol. 1986 Dec;61(12):790-7. No abstract available. Polish. PMID 3601483
- [Background] Aitio A. Effect of chrysene and carbon tetrachloride administration on rat hepatic microsomal monooxygenase and UDPglucuronosyltransferase activity. FEBS Lett. 1974 May 15;42(1):46-9. doi: 10.1016/0014-5793(74)80275-9. No abstract available. PMID 4211953
- [Background] Schmidt W, Merz WE, Lenhard V, Kubli F. Effects of crude and purified human chorionic gonadotropin on lymphocyte response. Gynecol Obstet Invest. 1981;12(3):132-40. doi: 10.1159/000299595. PMID 6453759
- [Background] Hall R, Ramaiah RS, Jones DT. General practitioner hospitals: coming or going? Br Med J (Clin Res Ed). 1984 Jun 2;288(6431):1691. doi: 10.1136/bmj.288.6431.1691-a. No abstract available. PMID 6426692
- [Background] Burke PM, Jancar J. Sensory and motor defect in severe mental subnormality. Ir J Med Sci. 1969 Oct;8(10):463-8. doi: 10.1007/BF02958617. No abstract available. PMID 5364076
- [Background] Clarke ED, Goulding KH, Wardman P. Nitroimidazoles as anaerobic electron acceptors for xanthine oxidase. Biochem Pharmacol. 1982 Oct 15;31(20):3237-42. doi: 10.1016/0006-2952(82)90556-1. PMID 6897358
- [Background] Heidrich HG, Strych W, Prehm P. Spontaneously released Plasmodium falciparum merozoites from culture possess glycoproteins. Z Parasitenkd. 1984;70(6):747-51. doi: 10.1007/BF00927127. PMID 6395533
- [Background] Miller TR. 100 cases of hemipelvectomy: a personal experience. Surg Clin North Am. 1974 Aug;54(4):905-13. doi: 10.1016/s0039-6109(16)40396-8. No abstract available. PMID 4428322
- [Background] Ladwa RA. Comparison of Syndol and paracetamol in the relief of dental pain. Br Dent J. 1981 Apr 7;150(7):187-8. doi: 10.1038/sj.bdj.4804571. No abstract available. PMID 6938217
- [Background] Hoskins IA, Hemming VG, Johnson TR, Winkel CA. Effects of alterations of zinc-to-phosphorus ratios and meconium content on group B Streptococcus growth in human amniotic fluid in vitro. Am J Obstet Gynecol. 1987 Sep;157(3):770-3. doi: 10.1016/s0002-9378(87)80047-9. PMID 3307431
- [Background] Kirsch WM, Stears JC. Radiographic identification and surgical excision of an epidermoid tumor of the pineal gland. Case report. J Neurosurg. 1970 Dec;33(6):708-13. doi: 10.3171/jns.1970.33.6.0708. No abstract available. PMID 5312639
- [Background] Agrawal HC, Fishman MA, Prensky AL. A possible block in the intermediary metabolism of glucose into proteins and lipids in the brains of undernourished rats. Lipids. 1971 Jun;6(6):431-3. doi: 10.1007/BF02531382. No abstract available. PMID 4330106
- [Background] Kanerud L, Hafstrom I. [Acute arthritis and subcutaneous fat necrosis as the first symptom of pancreatic cancer]. Lakartidningen. 1986 Feb 19;83(8):609-10. No abstract available. Swedish. PMID 3951286
- [Background] Ritter D. The need for risk assessment legislation. Risk Anal. 1988 Jun;8(2):169-70. doi: 10.1111/j.1539-6924.1988.tb01166.x. No abstract available. PMID 3413308
- [Background] Shah GN, Li J, Schneiderjohn P, Mooradian AD. Cloning and characterization of a complementary DNA for a thyroid hormone-responsive protein in mature rat cerebral tissue. Biochem J. 1997 Oct 15;327 ( Pt 2)(Pt 2):617-23. doi: 10.1042/bj3270617. PMID 9359437